CLINICAL TRIAL: NCT03487107
Title: A Multicenter, Single-arm, Open-label Study to Investigate the Efficacy and Safety of Yimitasvir Phosphate (DAG181)/Sofosbuvir(SOF) Combination for 12 Weeks in Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Phase 3 Study of Yimitasvir Phosphate Capsules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DDAG181PA-16-007
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Chronic HCV Infection
Keywords: Chronic Genotype 1 HCV Infection
MeSH Terms: interventions — Sofosbuvir; yimitasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOF 400 mg+DAG181 100 mg (Experimental): Patients with genotype 1 HCV infection without cirrhosis will receive SOF 400 mg+DAG181 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: DAG181

INTERVENTIONS:
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: sofosbuvir; Sovaldi®
Drug: DAG181 — 100 mg capsule administered orally once daily
  Other Names: Yimitasvir

SUMMARY:
The safety, tolerability and antiviral activity of DAG181/SOF in treatment-naive and treatment-experienced patients with chronic hepatitis C virus (HCV) genotype 1 infection.

DETAILED DESCRIPTION:
A phase III, multicenter, single-arm, open-label study to assess the safety, tolerability and antiviral activity of DAG181/SOF combination for 12 weeks in adult subjects with chronic genotype 1 HCV infection.

Approximately 360 HCV genotype 1 subjects without cirrhosis will be enrolled, treatment-experienced subjects are ≤20%. All subjects will receive DAG181 100 mg/ SOF 400 mg once daily for 12 weeks，with subsequent observation for 24 weeks after cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Male or female, age≥18 years;
3. A female subject is eligible to enter the study if it is confirmed that she is:

   1. Of non-childbearing potential (i.e., women who have had a hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal-women > 50 years of age with cessation (for≥12 months) of previously occurring menses), or
   2. Of childbearing potential (Women≤50 years of age with amenorrhea will be considered to be of childbearing potential). These women must have a negative serum pregnancy test at screening and negative urine pregnancy test at baseline before first dose of study drugs, and must use specific contraceptive methods from screening until 90 days after last dose of study drugs, such as complete abstinence from intercourse, vaginal ring, cervical cap or contraceptive diaphragm, IUD, etc.
4. All male subjects must agree to consistently and correctly use specific contraceptive methods with their female partner from screening until 90 days after last dose of study drugs(except for surgical sterilization), such as complete abstinence from intercourse, condom, and their female partner use contraceptives , vaginal ring , cervical cap or contraceptive diaphragm, IUD, etc;
5. Male subjects must agree to refrain from sperm donation from the date of screening until 90 days after the last dose of study drugs;
6. Confirmation of chronic HCV infection documented by either:

   1. A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit, or
   2. A liver biopsy performed prior to the Baseline/Day 1 visit with evidence of chronic HCV infection.
7. Serological detection of anti-HCV antibodies was positive at screening;
8. HCV RNA≥1×104 IU/mL at Screening;
9. HCV genotype 1a, 1b, or mixed 1a/1b at screening as determined by the Central Laboratory;
10. Classification as treatment naive or treatment experienced;
11. Absence of cirrhosis.

Exclusion Criteria:

1. Investigator assessed subjects have other clinically significant abnormalities (other than HCV), such as uncontrollable heart disease, respiratory, gastrointestinal, blood, nervous or other medical disorders, which may interfere with treatment, assessment, or compliance with the protocol;
2. Laboratory results outside of acceptable ranges at Screening;
3. HBsAg serology test results were positive at Screening;
4. HIV antibody test results were positive at Screening;
5. Prior exposure to approved or experimental HCV-specific direct-acting antiviral agent;
6. Pregnant female or male with pregnant female partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with sustained virologic response 12 weeks after discontinuation of therapy(SVR12) | Posttreatment Week 12
  SVR12 is defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after discontinuation of therapy
Safety and tolerability were evaluated based on adverse events | Up to posttreatment week 24
  Collecting all adverse events during the whole study

SECONDARY OUTCOMES:
Percentage of subjects with sustained virologic response 4 and 24 weeks after discontinuation of therapy (SVR4 and SVR24) | Posttreatment Weeks 4 and 24
  SVR4 and SVR24 were defined as HCV RNA < the lower limit of quantitation (LLOQ) at 4 and 24 weeks after discontinuation of therapy, respectively.
HCV RNA change from baseline | Up to posttreatment week 24
  the quantification of HCV RNA during and after treatment compared with baseline
Percentage of subjects with virologic failure | Up to posttreatment week 24
  1. On-treatment virologic failure:
     1. confirmed HCV RNA ≥ the lower limit of quantitation (LLOQ) after having previously had HCV RNA <the lower limit of quantitation (LLOQ) while on treatment;
     2. confirmed ≥ 1 log10 IU/mL increase in HCV RNA from nadir while on treatment;
     3. HCV RNA persistently ≥the lower limit of quantitation (LLOQ) through 8 weeks of treatment.
  2. Virologic relapse:
     1. Confirmed HCV RNA ≥the lower limit of quantitation (LLOQ) during the posttreatment period having achieved HCV RNA <the lower limit of quantitation (LLOQ) at last on-treatment visit.
Percentage of subjects with viral resistance to DAG181 and/or SOF | Up to posttreatment week 24
  Monitoring HCV virus resistance at baseline, during and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, Doctor, Study Chair — Peking University People's Hospital
Locations (35):
- China (35):
  - Beijing Ditan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University Science & Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The People's Liberation Army No.81 Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - The Fifth People's Hospital of Wuxi, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical Hospital, Xuzhou, Jiangsu
  - The Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No